CLINICAL TRIAL: NCT04785950
Title: An Observational, Prospective, Multicenter Study to Assess the Continuation Rates and User Acceptability of Bleeding Profile in First-time Users of Low-dose LNG-IUS
Brief Title: The Aim of This Study is to Estimate the Discontinuation Rate of Low-dose Levonorgestrel-releasing Intrauterine System Due to Self-reported Unacceptable Menstrual Bleeding Pattern in Spanish Women Who Are Using it for the First Time How Intrauterine System for Long Acting Contraception
Acronym: CORA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21279
Record Dates: First submitted 2021-02-04; First posted 2021-03-08 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Hormonal Intrauterine Contraception
Keywords: Intrauterine system (IUS); Levonorgestrel (LNG); Menstrual bleeding; Discontinuation of intrauterine systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with IUS: Women aged 18 to 35 years from Spain who chose to use any low-dose LNG-IUS marketed in Spain for the first time during routine clinical practice
  Interventions: Drug: Low-dose levonorgestrel intrauterine systems (LNG-IUS)

INTERVENTIONS:
Drug: Low-dose levonorgestrel intrauterine systems (LNG-IUS) — Any low-dose intrauterine system (IUS) marketed in Spain

SUMMARY:
Researchers are looking for better ways to help women prevent pregnancy. Every month, a woman's body prepares for pregnancy in a process called the menstrual cycle. When pregnancy does not happen, menstruation occurs. During menstruation, women lose blood and tissue from inside the womb. This bleeding can last for about 2 to 7 days.

Hormonal intrauterine contraception aims to help women prevent pregnancy by stopping the process of the menstrual cycle. Intrauterine means that the contraception is in the form of a device that is inserted into a woman's womb by her doctor. The device then releases the contraception into the womb.

Researchers have found that when women use hormonal contraception, the disruption to the menstrual cycle can cause changes to how often and for how long women will bleed. So, the researchers in this study want to learn more about the menstrual bleeding patterns of women in Spain who are using hormonal intrauterine contraception for the first time. In other words, In particular for the LNG-IUSs, irregular bleeding due to the local effect of levonorgestrel on the endometrium is common, particularly during the first 3 months of use, and it is of interest to know if this is a major reason why Spanish women discontinue this very effective method and what other factors may be associated with discontinuation. The researchers will then use this information to estimate how many women choose to stop using the contraception. The participants will be able to enroll in this study after requesting hormonal intrauterine contraception from their doctor. They will be women between the ages of 18 and 35 who have never used hormonal intrauterine contraception before.

The participants will visit the study site 3 times. On the first visit, they will receive the hormonal intrauterine contraception. The doctors will also check their health to make sure they can join the study. The participants will visit the study site again 4-12 weeks later, and one last time after 1 year of having the hormonal intrauterine contraception. During these visits, the doctors will ask the participants questions about any medical problems they have and if they want to continue using the contraception. Throughout the study, the participants will use a mobile app to track information about their menstrual bleeding and how they feel about it.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 35 years.
* Women who have freely chosen a low-dose LNG-IUS for the first time as contraceptive method and it has been successfully inserted previously to invite the woman to participate in the study.
* Women capable of reading and writing.
* Women who signed the informed consent form.
* Women who are not participating in an investigational program with interventions outside of routine clinical practice.
* Women without a mental illness and able to make decisions and follow instructions.
* Women without contraindications to a low-dose LNG-IUS according to the local marketing authorization.
* Women without concomitant medications that may lead to changes in the bleeding pattern (e.g. antiplatelet and/or anticoagulants).

Exclusion Criteria:

* None

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adult women from Spain
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Percentage of women who discontinue the use of low-dose LNG-IUS due to the unacceptability of their menstrual bleeding pattern | Up to 12 months

SECONDARY OUTCOMES:
Percentage of women who discontinued lowdose LNG-IUS due to other reasons | At final visit (up to 12 months)
Women's perception of the amount of information received during preinsertion counselling about the potential changes in menstrual bleeding pattern after lowdose LNG-IUS insertion | At final visit (up to 12 months)
  Did you received information during pre-insertion counselling about the potential changes in menstrual bleeding pattern after low-dose LNG-IUS insertion?
  * A lot
  * Quite a lot
  * A moderate amount
  * Relative little
  * Very little
Potential correlation of women's perception on pre-insertion counselling with overall satisfaction with menstrual bleeding pattern | At final visit (up to 12 months)
Usage of the mobile apps to support menstrual tracking (regularly, sporadically, never) | At initial visit, follow-up and final visit (up to 12 months)
Overall satisfaction with the menstrual app (very satisfied; satisfied; neither satisfied nor dissatisfied; dissatisfied; very dissatisfied) | At initial visit, follow-up and final visit (up to 12 months)
Correlation between the use of a menstrual app and discontinuation | At initial visit, follow-up and final visit (up to 12 months)
Correlation between the use of a menstrual app and overall satisfaction with menstrual bleeding pattern | At initial visit, follow-up and final visit (up to 12 months)
Size of uterine cavity | At initial visit (Day 0)
Menstrual bleeding pattern with 8 parameters | Up to 12 months
  8 Parameters:
  * Presence/absence of menstrual bleeding
  * Frequency: frequent: <24 days; normal: 24-38 days; infrequent: >38 days
  * Regularity of withdrawal bleeding: regular, one bleeding episode per cycle; irregular, all those cycles that are not regular
  * Duration: long: >8 days; normal: 4-8 days; short: <4 days
  * Quantity: 10 cm visual analogue scale (VAS) (on the left "absence of bleeding"; on the right "worst imaginable bleeding")
  * Menstrual pain: 10 cm VAS (on the left "no pain"; on the right "worst imaginable pain"
  * Presence/absence of intermenstrual vaginal bleeding or spotting: yes; no
  * Interference in daily activities: not at all; mildly; moderately; severely
Change of menstrual bleeding pattern with 8 parameters between baseline and 4 to12 weeks / final visit | Up to 12 months
  8 Parameters:
  * Presence/absence of menstrual bleeding
  * Frequency: frequent: <24 days; normal: 24-38 days; infrequent: >38 days
  * Regularity of withdrawal bleeding: regular, one bleeding episode per cycle; irregular, all those cycles that are not regular
  * Duration: long: >8 days; normal: 4-8 days; short: <4 days
  * Quantity: 10 cm visual analogue scale (VAS) (on the left "absence of bleeding"; on the right "worst imaginable bleeding")
  * Menstrual pain: 10 cm VAS (on the left "no pain"; on the right "worst imaginable pain"
  * Presence/absence of intermenstrual vaginal bleeding or spotting: yes; no
  * Interference in daily activities: not at all; mildly; moderately; severely
Correlation between uterine cavity size and menstrual bleeding pattern | Up to 12 months
Overall satisfaction with menstrual bleeding pattern assessed on a 5-point Likert scale (Very satisfied; Satisfied; Neither satisfied nor dissatisfied; Dissatisfied) | At baseline, at the follow-up visit and at the final visit (up to 12 months)
Change in satisfaction with menstrual bleeding pattern assessed on a 5-point Likert scale (Very satisfied; Satisfied; Neither satisfied nor dissatisfied; Dissatisfied) between baseline and 4-12 weeks / final visit | At baseline, at the follow-up visit and at the final visit (up to 12 months)
Correlation between overall satisfaction with menstrual bleeding and the menstrual bleeding pattern | At baseline, at the follow-up visit and at the final visit (up to 12 months)
Percentage of women that would recommend the use of low-dose LNG-IUS to a friend | At final visit (up to 12 months)
Days up to discontinuation day | at the follow-up visit and at the final visit (up to 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.